CLINICAL TRIAL: NCT03998943
Title: NOCTURNAL PAIN After Knee Arthroplasty : Incidence and Risk Factor: an Observational Study
Acronym: NOCTURN-PAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/17AVR/182
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis; Pain, Postoperative; Prosthesis (Internal) Complications; Nocturnal Frequency
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative; Nocturia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In prosthetic knee surgery, there is a certain number of patients with post-operative nocturnal pain. The purpose of our study is to determine the impact of this problem and to better understand its risk factors.

DETAILED DESCRIPTION:
In prosthetic knee surgery, there is a certain number of patients with post-operative nocturnal pain.

The purpose of our study is to determine the impact of this problem and to better understand its risk factors.

This is a poorly studied issue and the study could better detect, evaluate and treat painful patients after knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective primary Total knee arthroplasty or unicompartmental knee arthroplasty due to knee joint osteoarthritis
* Older than 18 years
* Willing and able to complete pre and postoperative surveys

Exclusion Criteria:

* History of drug abuse
* Previous knee arthroplasty
* Mental disorders
* Rheumatoid arthritis
* Chronic renal disease
* Chronic hematological diseases (sickle cell disease, haemochromatosis...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients undergoing elective primary Total knee arthroplasty or unicompartimental knee arthroplasty due to knee joint osteoarthritis coming to elective surgery at Cliniques universitaires Saint-Luc, Brussels
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
nocturnal pain | from day 1 of surgery until 1 year post surgery
  response to question (yes-no) "Does the pain in the operated knee wake you up at night or prevent you from sleeping?"

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Thienpont, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No